CLINICAL TRIAL: NCT01965314
Title: Randomised Control Trial to Determine the Effect of Simulation Based Training on Initial Performance of Ultrasound Guided Axillary Brachial Plexus Blockade in a Clinical Setting
Brief Title: A Trial to Determine the Effect of Simulation Based Training on Initial Performance of Ultrasound Guided Axillary Brachial Plexus Blockade in a Clinical Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. The simulator lacked the fidelity required to meet training needs of the novices, 2. Recruitment of novice anesthetists more difficult than anticipated
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Owen O'Sullivan, Research Fellow, Department of Anaesthesia, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Haystack USgABPB sim-training
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesiology Training
Keywords: ultrasound guided regional anaesthesia; upper limb surgery; ultrasound guided axillary brachial plexus blockade

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Training Group (Placebo Comparator): These subjects will be offered multimodal training. This will be comprised of demonstration by suitably trained individuals of relevant anatomy using pre-existing cadaveric samples, performing ultrasound scans of the relevant areas on volunteers under expert supervision, and the practice of needle insertion under ultrasound-guidance using commonly used tissue phantoms (turkey breasts).
  Interventions: Other: Traditional training
- Simulation Training Group (Active Comparator): In addition to traditional training the SG group will participate in a period of simulator based training. Following initial familiarization with the simulator these participants will identify relevant structures and follow their course in the virtual arm. They will insert a virtual needle into the virtual environment and advance it using an in-plane technique towards various target structures. They will be given immediate directed computer generated feedback and offered the opportunity for repetitive, deliberate practice. The simulator, which these participants will use, will comprise of a PHANTOM Desktop (http://www.sensable.com/), an haptic immersive workbench and the H3D API (http://www.sensegraphics.se/). The SG subject will scan and perform procedure specific tasks on a virtual arm. Training will continue until they reach proficiency levels set by experts using the same simulator.
  Interventions: Other: Simulation based training; Other: Traditional training

INTERVENTIONS:
Other: Simulation based training — In addition to traditional training (as delivered to participants in the Traditional Training Group), participants in the Simulation Training Group will receive the following:- Following initial familiarization with the simulator SG participants will identify relevant structures and follow their course in the virtual arm. They will insert a virtual needle into the virtual environment and advance it using an in-plane technique towards various target structures. They will be given immediate directed computer generated feedback and offered the opportunity for repetitive, deliberate practice. The simulator, which SG participants will use, will comprise of a PHANTOM Desktop (http://www.sensable.com/), an haptic immersive workbench and the H3D API (http://www.sensegraphics.se/). The SG subject will scan and perform procedure specific tasks on a virtual arm. Training will continue until they reach proficiency levels set by experts using the same device
  Arms: Simulation Training Group
Other: Traditional training — Subjects will be offered standardized multimodal training. This will be comprised of demonstration by suitably trained individuals of relevant anatomy using pre-existing cadaveric samples, performing ultrasound scans of the relevant areas on volunteers under expert supervision, and the practice of needle insertion under ultrasound-guidance using commonly used tissue phantoms (turkey breasts).

SUMMARY:
Investigators hypothesize that virtual reality based training offers an additional learning benefit over standard training (using cadaveric dissection and human volunteers) in preparing novice anaesthetists to perform their first Ultrasound guided Axillary Brachial Plexus Blockade (USgABPB) in the clinical setting.

Investigators hope that this body of work will aid the development of a visuo-haptic simulator used to improved training of doctors in performing USgABPB. Ultimately any patient having this procedure carried out in the future should benefit. In particular it will avoid the need for novice trainees to practice new techniques on patients.

DETAILED DESCRIPTION:
Ultrasound guided axillary brachial plexus blockade (USgABPB) is a commonly performed medical procedure which enables the performance of surgery on the upper limb without general anaesthesia. Its competent performance entails complex, simultaneous interactions between three processes. These are active management of the patient, acquisition and interpretation of ultrasound images, and the placement a needle tip close to specific nerves to facilitate deposition of local anaesthetic. Currently, the procedure is taught using two-dimensional drawings, cadaveric specimens, videos, 3D animations, live demonstrations, and/or supervised clinical practice. Simulated practice, using tofu-based or animal models, have been used to bridge the gap from knowledge to clinical performance. Training in medical procedural skills is currently undergoing important change. Factors including altered patient expectations and the European Working Time Directive (2000/34/EC amending Directive 93/104/EC) limit the number of clinical learning opportunities available to trainees. These changes are likely to decrease particularly the number of opportunities for trainees to learn and practice procedural skills in a clinical setting. The traditional Halstedian apprenticeship model of medical training is being challenged. In this model, training is associated with progressively less supervision as part of progressive independence. "See one, do one" is no longer an appropriate method for teaching procedural skills because patients are necessarily exposed to inexperienced practitioners. This model requires a large investment of time by both trainer and trainee in the clinical environment. Its application decreases the efficiency of operating room activity. These circumstances pose medical trainers and training bodies with a dilemma, a decrease in the number of individual opportunities implies that the total duration of training should increase or a lesser level of competence accepted at completion of training

Simulation has been used widely for training in and assessment of medical procedural skills. Applied to essential anaesthetic skills, simulation may be more efficient than the apprenticeship approach. This may offer a partial solution to the problem of limited clinical learning opportunities for USgPNB. Simulated practice with formative feedback has been shown to be of benefit in the rapid acquisition of basic ultrasound skills by inexperienced clinicians. Ultimately, the purpose of simulated practice of medical procedures is to enhance clinical performance. One proven important role for simulation is to prepare novice clinicians to bridge the gap between acquiring knowledge and initial clinical performance. Significantly, the Food and Drug Administration (FDA) has recently mandated that clinicians who perform carotid stenting using a particular stent should train to a defined level of proficiency on a simulator before they perform the procedure on a patient.

With institutional ethical approval and having obtained written informed consent from participants (patients and anaesthetists) 20 College of Anaesthetists (RCSI) affiliated trainees who have no experience of performing ultrasound guided regional anaesthesia will be recruited. Participating anaesthetists will provide baseline personal data including previous experience with peripheral nerve blockade and simulators, using a web-based collection facility (www.surveymonkey.com or similar). They will perform baseline psychomotor tests prior to beginning training. Baseline visuo-spatial ability will be assessed using the card rotation, cube comparison, and map planning tests (Educational Testing Service) or similar. Psychomotor ability will be assessed using a grooved pegboard (Lafayette Instruments, Lafayette, IN) or similar. All participating anaesthetists will receive standardized two hour didactic training encompassing relevant anatomy, ultrasound (physics, function and interpretation), pharmacology of relevant agents, indications/ contraindications of the block and complications of the procedure. Participants will be taught to perform USgABPB using a technique as described in Appendix IV and V of 'The American Society of Regional Anesthesia and Pain Medicine and the European Society of Regional Anaesthesia and Pain Therapy Joint Committee Recommendations for Education and Training in Ultrasound-Guided Regional Anesthesia'. This technique uses a transverse (or short-axis) view, on ultrasound imaging, of the axillary brachial plexus and axillary blood vessels. The needle is inserted in a sterile fashion using an 'in-plane' approach, that is, the needle shaft and tip will remain visible on ultrasound view throughout it course towards the relevant nerves. Following this initial period of common training subjects will be randomly allocated (using computer generated random numbers) to one of two groups of equal size for additional training which will occur in parallel over a two hour period, namely a simulator trained group (SG) or a control group (CG). Following the educational intervention all subjects will be asked to give written feedback on the content and delivery of the session.

Traditional training TG subjects will be offered multimodal training. This will be comprised of demonstration by suitably trained individuals of relevant anatomy using pre-existing cadaveric samples, performing ultrasound scans of the relevant areas on volunteers under expert supervision, and the practice of needle insertion under ultrasound-guidance using commonly used tissue phantoms (turkey breasts). All ultrasound examinations performed on volunteers or during the clinical performance on patients will use a Sonosite M Turbo (or similar device) with a 7-12 MHz 38mm linear probe. This training session will last two hours.

Simulator training In addition to traditional training the SG group will participate in a period of simulator based training. Following initial familiarization with the simulator SG participants will identify relevant structures and follow their course in the virtual arm. They will insert a virtual needle into the virtual environment and advance it using an in-plane technique towards various target structures. They will be given immediate directed feedback by an expert and offered the opportunity for repetitive, deliberate practice. The simulator, which SG participants will use, will comprise of a PHANTOM Desktop (http://www.sensable.com/), an haptic immersive workbench and the H3D API (http://www.sensegraphics.se/). The SG subject will scan and perform procedure specific tasks on a virtual arm. The model of the arm will be informed using MRI or ultrasound supervolume DICOM datasets. This training session will last two hours.

Assessment Within two weeks of the educational intervention all participants' first clinical performance of an ultrasound guided nerve block, specifically an ultrasound guided axillary brachial plexus blockade, will be video recorded for subsequent analysis by two experts in UGRA. Patients involved will require anaesthesia for forearm/wrist/hand surgery where USgABPB would ordinarily be offered as standard care. Subsequent care of the patient may include general anaesthesia, as clinically indicated. Intravenous sedation will be offered and administered as clinically indicated (Midazolam up to a maximum of 0.05mg/kg).

Subjects will perform the procedure, using an in-plane approach and short-axis view (see above), in the presence of a supervising trainer, blinded to training group, who is available to intervene if required, for patient safety, or requested by the subjects themselves. Patients involved will also be blinded to subject allocation. Using a video recording device Sony Handycam HDR-XR520VE, or similar, the performance of a clinician indicated USgABPB for a scheduled operation on patients will be recorded. The video-taping will target primarily the anaesthetist performing the clinically indicated ultrasound guided regional anaesthetic technique in the usual fashion at Cork University Hospital. The recording will proceed in a manner aimed to conceal the identity of the patient and maintain confidentiality. All efforts will be taken to ensure the recording will not include images of the patients face. For the purpose of blinding, a similar effort will be made conceal the identity of the anaesthetists performing the block by avoiding shots of their faces. The recording will include a pan shot of the setup of the room the block will take place in. This will indicate the location of the patient, the ultrasound machine, the trolley with the sterile equipment required, the assistant, the monitor, the emergency drugs, and the anaesthetist performing the block. Before commencing the block the camera will be fixed in position focusing on the axilla, with needle insertion site, ultrasound probe and the movements of the anaesthetist's hands recorded. The acquired ultrasound image will be recorded concurrently. After expert assessment of trainee performance and completion of the dataset all recorded video will be destroyed.

For the purpose of the study the subjects will be give some specific directions.

1. Position the patient and equipment appropriately.
2. They will be asked to perform a pre-procedure ultrasonic survey of the relevant area, specifically identifying the four relevant nerves (musculocutaneous, radial, median, and ulnar).
3. Perform a sterile four nerve ultrasound-guided axillary brachial plexus block, utilizing a single skin entry point (where possible), short axis view of the brachial plexus, and needle in-plane approach.
4. They will be asked to demonstrate the effectiveness of the blockade.

Following the recorded performance of the procedure the subjects will be asked to complete a written questionnaire indicating their confidence in performing the procedure and their perception of the influence of external stressors (including the presence of a camera).

ELIGIBILITY:
Patients

Inclusion Criteria:

* ASA grades I and II
* Age 18-80 years
* Capacity to consent
* Already consented for ultrasound guided axillary brachial plexus blockade
* Body Mass index 20 - 26

Exclusion Criteria:

* Parameters outside inclusion criteria
* Contraindication to regional anaesthesia
* Language barrier
* Psychiatric history
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
positive total of procedural checklist items | As assessed by retrospective video analysis of procedure (from patient positioning to assessment of adequacy of block) by two blinded experts (within 6 months of procedure)
  Yes or No which of the following elements were performed
  1. Conducts clear pre-procedural consultation with patient
  2. Obtains informed consent
  3. Secures IV Access
  4. Applies appropriate monitoring
  5. Prepares equipment and emergency drugs appropriate for standard regional anaesthesia procedures
  6. Selects appropriate local anaesthetic agents
  7. Works with trained assistant
  8. Prepares sterile Regional Trolley
  9. Selects linear broadband transducer with 5-13MHz frequency
  10. Uses US coupling gel and sterile cover
  11. Uses 50 mm needle
  12. Positions patient semi recumbent with head supported for comfort
  13. Positions operative arm in-90° abduction and externally rotates and supports in comfortable position
  14. Elevates bed position to appropriate level
  15. Positions the performer and US screen on the operative side with the screen cephalad to the trolley etc...(limited by character count)

SECONDARY OUTCOMES:
procedural times | (During procedure) From patient and equipment positioning to assessment of adequacy of block
number of needle passes | during the procedure
  A numerical count of the number of times the needle is inserted ands removed during performance of the procedure.
block success | within 15 mins of the procedure
  as defined by sensory & motor blockade in the distribution of all four relevant nerves demonstrated within 15 minutes of USgABPB
participating anaesthetist confidence levels | immediately following performance of the USgABPB (within 30 minutes)
  measured on a ten point verbal rating scale, on completion of assessment of the block - "How confident were you in performing the block?"
patient satisfaction measure | prior to discharge from the post anaesthesia care unit (recovery room) - (not more than 2 hours following completion of surgical procedure requiring anaesthesia)
  measured on a ten point verbal rating scale, on discharge from recovery "How satisfied were you with the block?"
global rating scale (GRS) scores | On retrospective video analysis of procedure (from patient positioning to assessment of adequacy of block)by blinded observers (within 6 months of procedure)
  Global Rating Scale
  Indicate on a continuous scale of 0-10 the manner in which the learner displays the following qualities:
  1. Good clinical judgement including patient selection
  2. Establishes and maintains rapport with the patient
  3. Confident and reassuring manner
  4. Patient, friendly and understanding manner
  5. Good communication skills with patient and team
  6. Organised, disciplined, plans ahead and uses time efficiently
  7. Attention to sterile technique
  8. Demonstrates ergonomics of movement and dexterity
  9. Checks hand/probe/needle position intermittently
  10. Gentle needle technique
  11. Safety conscious
  12. Attentive to patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: George Shorten, PhD, Principal Investigator — Cork University Hospital & University College Cork
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

REFERENCES:
- [Derived] O'Sullivan O, Iohom G, O'Donnell BD, Shorten GD. The effect of simulation-based training on initial performance of ultrasound-guided axillary brachial plexus blockade in a clinical setting - a pilot study. BMC Anesthesiol. 2014 Nov 26;14:110. doi: 10.1186/1471-2253-14-110. eCollection 2014. PMID 25844062